CLINICAL TRIAL: NCT03739398
Title: A Study on the Effectiveness and Safety Evaluation of Combination Therapy With 1,927nm Thulium Laser and Fractional Microneedle Radiofrequency Equipment for Improvement of Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2018-0045
Record Dates: First submitted 2018-10-30; First posted 2018-11-13 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Wrinkle

STUDY DESIGN:
Intervention Model Description: LUTRONIC GENIUS Laser is performed on one side and LASEMD Laser is performed on the other. LUTRONIC GENIUS Laser is performed on the other side without energy irradiation. Laser treatment is performed after application of EMLA cream (2.5% lidocaine 2.5% and prilocaine 2.5%) for 30 minutes or more before local anesthesia.
  Measurement of hydration, transepidermal water loss, skin pigmentation, redness, and elasticity were performed using a corneometer, a vapometer, a mexameter, and a cutometer before the procedure and on the 7th day after the first operation and 3 months after the last operation. Using an Antera 3D® camera, the skin texture, wrinkles, pores, volume of depressions / elevations, skin color, redness and pigmentation were measured. The change of skin surface and extent of wrinkle were measured using a visuometer, a high-resolution camera.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUTRONIC GENUS laser with LASEMD laser (Experimental)
  Interventions: Device: LUTRONIC GENUS laser(Fractional Microneedle Radiofrequency(FMR))
- LUTRONIC GENUS laser without LASEMD laser (Active Comparator)
  Interventions: Device: LASEMED laser(The Thulium laser with 1,927nm wavelength)

INTERVENTIONS:
Device: LUTRONIC GENUS laser(Fractional Microneedle Radiofrequency(FMR)) — 1. LUTRONIC GENUS laser(Fractional Microneedle Radiofrequency(FMR)) : Fractional Microneedle Radiofrequency (FMR) equipment is a device that penetrates the epidermis and irradiates the high frequency by entering the dermis. The generated radiofrequency transfers heat energy and induces thermal denaturation in the surrounding tissue. Using this principle, FMR equipment is being used as a very effective treatment for scarring, enlarged pores, hyperhidrosis as well as wrinkles. Unlike conventional treatments, FMR equipment has the advantage of a short recovery time after treatment because it minimizes damage to the epidermis because the insulated microspheres penetrate the skin and generate high frequency only at the end of the microspheres.
  Arms: LUTRONIC GENUS laser with LASEMD laser
Device: LASEMED laser(The Thulium laser with 1,927nm wavelength) — 2. LASEMD laser(The Thulium laser with 1,927nm wavelength) The Thulium laser with 1,927nm wavelength is a device that effectively removes various skin diseases present in the epidermis while minimizing the side effects such as scarring and pigmentation because it induces thermal damage to the only skin surface compared to conventional laser equipment. In recent years, not only skin lesions on the epidermis but also pigment disease and wrinkles have been reported to have a good effect.
  In this study, we investigated the effect and stability of combined treatment of Thulium laser with 1,927nm wavelength in addition to FMR equipment which has already proven to be effective in improving skin aging.
  Arms: LUTRONIC GENUS laser without LASEMD laser

SUMMARY:
Fractional Microneedle Radiofrequency (FMR) equipment is a device that penetrates the epidermis and irradiates the high frequency by entering the dermis. The generated radiofrequency transfers heat energy and induces thermal denaturation in the surrounding tissue.

DETAILED DESCRIPTION:
Using this principle, FMR equipment is being used as a very effective treatment for scarring, enlarged pores, hyperhidrosis as well as wrinkles. Unlike conventional treatments, FMR equipment has the advantage of a short recovery time after treatment because it minimizes damage to the epidermis because the insulated microspheres penetrate the skin and generate high frequency only at the end of the microspheres.

The Thulium laser with 1,927nm wavelength is a device that effectively removes various skin diseases present in the epidermis while minimizing the side effects such as scarring and pigmentation because it induces thermal damage to the only skin surface compared to conventional laser equipment. In recent years, not only skin lesions on the epidermis but also pigment disease and wrinkles have been reported to have a good effect.

In this study, investigator investigated the effect and stability of combined treatment of Thulium laser with 1,927nm wavelength in addition to FMR equipment which has already proven to be effective in improving skin aging.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy normal adults between 45 and 65 years of age
2. Subjects with moderate to severe wrinkles based on the Investigator's global assessment of lateral canthal line severity rating
3. Subjects who have voluntarily signed a written consent before
4. Subjects who can follow up during the trial
5. Subjects who have agreed to cease all dermatological treatment or treatment, including improvement of neck and face wrinkles, during this trial

Exclusion Criteria:

1. If subjects do not want it or do not fill out a consent form
2. If subjects are allergic to local anesthetics (lidocaine)
3. Subjects who are Pregnant or lactating
4. Subjects who are deemed to be inadequate as subjects by the clinical investigator for the following patients or other pathologies 1) If the site of treatment has infectious or inflammatory skin disease 2) If the site of treatment has melasma or other pigmented dermatologic disease 3) If subjects have keloid disease, collagen, or elastic fiber disease 4) If subjects have chronic wasting disease (asthma, diabetes, etc.) 5) If subjects are taking anticoagulants and are at risk of bleeding 6) If subjects have an autoimmune disease 7) Subjects with psychiatric problems 8) Acute patients
5. Others in addition to the above items, if it is deemed difficult for clinical practice to be conducted at the discretion of the clinical trial manager (including illiteracy and other foreigners exclusion)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Skin roughness | immediately before the procedure to three months after last procedure
  The roughness and wrinkle of the skin corresponding to the wrinkles of the outer eyelid
wrinkle | immediately before the procedure to three months after last procedure
  the wrinkle of glabella were measured using an Antera 3D camera and compared

SECONDARY OUTCOMES:
Transepidermal water loss | immediately before the procedure to three months after last procedure
Description of overall manifestation by clinical photo and visiometer | immediately before the procedure to three months after last procedure
  pigmentation, erythema, scaliness will be checked by photo and visiometer
Patients' subjective Treatment Satisfaction of the degree of skin aging improvement, wrinkles, pores, skin color, skin elasticity, skin dryness | immediately before the procedure to three months after last procedure
  (0 : Not satisfied, 1 : Somewhat satisfied, 2 : Satisfied, 3: Very satisfied)
Evaluation of researchers' skin improvement | immediately before the procedure to three months after last procedure
  (0 : Not improved, 1 : 1 ~ 25% improvement, 2 : 26 ~ 50% improvement, 3: 51 ~ 75% improvement, 4: More than 76% improvement)
Change of investigator's global assessment of lateral canthal line severity rating | immediately before the procedure to three months after last procedure
  ( 0: Absent, 1: minimal, 2 : mild, 3: moderate, 4: severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Severance Hospital, Cutaneous Biology Research Institute, Yonsei University College of Medicine, Seoul, South Korea